CLINICAL TRIAL: NCT03005535
Title: Randomised Clinical Trial to Assess the Medium-term Effect of 30 g/Day of a Vitaminised Corn Oil or Olive Oil, on Lipid Parameters, Vascular Risk Markers Blood Pressure and Endothelial Function, in Moderately Hypercholesterolemic Subjects
Brief Title: Effects of Corn Oil Plus Vitamin E and B6 on LIpids, PcSk9 and Endothelial Function
Acronym: ECLIPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Chief Internal Medicine Unit, University of Bologna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ECLIPSE_2016
Record Dates: First submitted 2016-12-05; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitaminized corn oil (Active Comparator): Vitaminized corn oil (plus B6 and E vitamins), 30 g per day, per 8 weeks, with meals (15 g per meal)
  Interventions: Other: Vitaminized corn oil
- Olive oil (Placebo Comparator): Olive oil (not extra-virgin), 30 g per day, per 8 weeks, with meals (15 g per meal)
  Interventions: Other: Olive oil

INTERVENTIONS:
Other: Vitaminized corn oil — Oil consumption at the two main meals, lunch and dinner (15gx2 per day)
  Arms: Vitaminized corn oil
Other: Olive oil — Oil consumption at the two main meals, lunch and dinner (15gx2 per day)
  Arms: Olive oil

SUMMARY:
This will be a randomized clinical trial carried out on subjects with suboptimal control of cholesterolemia who will consume 30 g per day of a vitaminized corn oil (plus B6 and E vitamins), in order to evaluate the effects on lipid profile, endothelial function and PCSK9

DETAILED DESCRIPTION:
In order to assess the mid term effects of vitaminized corn oil on endothelial function and on early markers of functional damage of the arterial wall, moderately hypercholesterolemic subjects will be supplemented for 8 weeks with 30 g/day of both a vitaminized corn oil (plus B6 and E vitamins) or olive oil. The two intervention periods will be spaced by a 4 week washout period.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol between 200 and 280 mg/dL and/or LDL cholesterol between 130 and 190 mg/dL
* Triglycerides lower than 200 mg/dL
* Cardiovascular risk at 10 years lower than 10%
* Informed consent

Exclusion Criteria:

* Secundary prevention for cardiovascular diseases
* BMI higher than 30
* Assumption of lipid lowering drug or supplement
* Alcohol abuse
* Alterations in thyroid, liver or kidney functions, muscle diseases

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Endothelial function (measured by Endocheck) change from the baseline to the end of the intervention period | At the beginning and after 8 weeks of both intervention periods (up to 24 weeks)
12 hour fasting lipid profile change from the baseline to the end of the intervention period | At the first visit (run-in) at the beginning, after 4 and 8 weeks of both intervention periods (up to 24 weeks)
PCSK9 levels change from the baseline to the end of the intervention period | At the beginning and after 8 weeks of both intervention periods (up to 24 weeks)

SECONDARY OUTCOMES:
Inflammatory markers (high sensitivity C reactive protein hs-PCR, malondialdehyde MDA, homocysteine) change from the baseline to the end of the intervention period | At the beginning and after 8 weeks of both intervention periods (up to 24 weeks)
Blood pressure change from the baseline to the end of the intervention period | 6 months
Fatty acid profile of whole blood total lipids change from the baseline to the end of the intervention period | At the beginning and after 8 weeks of both intervention periods (up to 24 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Yes